CLINICAL TRIAL: NCT03287037
Title: To Investigate the Effect of Transcranial Direct Current Stimulation (tDCS) on Depressive Symptoms, Neurocognitive Function and Heart Rate Variability in Unipolar Depression and Bipolar Depression
Brief Title: The Effects of tDCS on Depressive Symptoms,Neurocognitive Function and HRV in Unipolar Depression and Bipolar Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Hsin-An Chang, MD, Head of Laboratory of Psychophysiology, Department of Psychiatry, Principal Investigator, Attending Psychiatrist, Assistant Professor, Tri-Service General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2-103-03-002-1
Record Dates: First submitted 2017-09-14; First posted 2017-09-19 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Depressive Disorder, Major; Depression, Bipolar; Electricity; Effects
Keywords: Unipolar depression; bipolar depression; Transcranial direct current stimulation
MeSH Terms: conditions — Depressive Disorder, Major; Bipolar Disorder; Depressive Disorder

STUDY DESIGN:
Intervention Model Description: Sixty patients with unipolar depression (major depressive disorder) and 60 with bipolar depression were treated with 10 sessions of tDCS.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- tDCS over DLPFC (Experimental): Direct current (DC) generated by a DC stimulator (Eldith DC stimulator: www. neuroconn.de/dc-stimulator_plus_en/) was bilaterally delivered through a pair of saline-soaked surface sponge electrodes (35 cm2). The anodal electrode was placed over the left dorsolateral prefrontal cortex (F3, International EEG System 10-20) and cathode electrode over F4. Stimulation was applied at an intensity of 2 mA for 20 min, twice-daily on 5 consecutive weekdays. The twice daily sessions were separated by at least 3 hours.
  Interventions: Device: tDCS over DLPFC

INTERVENTIONS:
Device: tDCS over DLPFC — We applied tDCS over dorsolateral prefrontal cortex (DLPFC) for these depressed patients. Direct current (DC) generated by a DC stimulator (Eldith DC stimulator: www. neuroconn.de/dc-stimulator_plus_en/) was bilaterally delivered through a pair of saline-soaked surface sponge electrodes (35 cm2). The anodal electrode was placed over the left dorsolateral prefrontal cortex (F3, International EEG System 10-20) and cathode electrode over F4. Stimulation was applied at an intensity of 2 mA for 20 min, twice-daily on 5 consecutive weekdays. The twice daily sessions were separated by at least 3 hours. All patients were maintained on their treatment throughout the study period.

SUMMARY:
The study aimed to investigate whether transcranial direct current stimulation could improve depressive symptoms, neurocognitive function and modulate heart rate variability in unipolar and bipolar depression.

DETAILED DESCRIPTION:
Background

Transcranial direct current stimulation encompasses the induction of a relatively weak constant current flow through the cerebral cortex via scalp electrodes . Dependent on stimulation polarity, this results in a modulation of cortical excitability and spontaneous neural activity. The technique was established in the 1950s and 1960s primarily in animals. In these early studies it was shown that subthreshold DC stimulation increases spontaneous neuronal activity if the anode is placed above or within the cortex, while exposure to cathodal polarity results in reduced activity. This is caused by a subthreshold membrane depolarization by anodal and a hyperpolarization by cathodal stimulation. It was demonstrated in humans that the after-effects of tDCS depend on modifications of NMDA receptor-efficacy. The after-effects of tDCS are blocked by the NMDA receptor antagonist dextromethorphan, and prolonged by the partial NMDA receptor-agonist D-cycloserine. This tDCS polarity-dependent alteration of NMDA receptor function seems to be initiated by the respective membrane potential shift and probably by the accompanying cortical activity modification,because it is prevented by the sodium channel blocker carbamazepine. Intraneuronal calcium concentration also contributes, because calcium channel antagonists eliminate the excitability-enhancing after-effects of anodal tDCS. Recently, tDCS has been reported to be a novel, non-invasive and safe therapeutic tool to treat neuropsychiatric disorders including depression. This therapeutic tool has been reported to show promising effect in treating unipolar and bipolar depression. However, the sample sizes have been small. Further work is needed to see if these early promising studies replicate. Much evidence has indicated that patients with depression show hypoactivity over left dorsolateral prefrontal cortex (DLPFC) and hyperactivity over right DLPFC. We therefore hypothesize that tDCS over DLPFC with anode placed at left DLPFC and cathode placed at right DLPFC would reduce depressive symptoms in patients with unipolar depression and bipolar depression.

The study aimed to investigate whether tDCS over DLPFC could modify depressive symptoms, neurocognitive function and heart rate variability of unipolar and bipolar depression.

Study design: open-label study.

Participants: 60 patients with unipolar depression and 60 with bipolar depression.

Others: see Arms and Interventions, Eligibility Criteria or Outcome Measures.

ELIGIBILITY:
Inclusion Criteria:

Patients who met DSM-IV-TR criteria for major depressive disorder and bipolar depression and had moderate to severe depression severity (HAM-D score more than 17) were included in the study.

Exclusion Criteria:

1. pregnancy or breastfeeding.
2. having epilepsy, severe physical illness, any current psychiatric comorbidity or history of substance dependence.
3. having contraindications for transcranial electrical/magnetic stimulation.
4. having intracranial metal foreign bodies.
5. having a history of intracranial neoplasms or surgery, or a history of severe head injuries or cerebrovascular diseases.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2019-09-06 (Actual); Study Completion 2019-09-06 (Actual)

PRIMARY OUTCOMES:
Changes from baseline score of Hamilton Depression Rating Scale (HAM-D) at the timepoint immediately after tDCS, at one week and one month after tDCS | One month
  Depression severity

SECONDARY OUTCOMES:
Changes from baseline score of Young Mania Rating Scale (YMRS) at the timepoint immediately after tDCS, at one week and one month after tDCS | One month
  Hypomania/mania severity
Changes from baseline score of Hamilton Anxiety Rating Scale (HAM-A) at the timepoint immediately after tDCS, at one week and one month after tDCS | One month
  Anxiety severity.
Changes from basline heart rate variability (HRV) at the timepoint immediately after tDCS, at one week and one month after tDCS | One month
  Index of autonomic functioning.
Changes from baseline results of continuous performance test (CPT) at the timepoint immediately after tDCS, at one week and one month after tDCS | One month
  Performance of prefrontal-mediated task.

CONTACTS AND LOCATIONS:
Overall Officials: Hsin-An Chang, M.D., Principal Investigator — Tri-Service General Hospital, National Defense Medical Center
Locations (1):
- Tri-service general hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lin YY, Chang CC, Huang CC, Tzeng NS, Kao YC, Chang HA. Efficacy and neurophysiological predictors of treatment response of adjunct bifrontal transcranial direct current stimulation (tDCS) in treating unipolar and bipolar depression. J Affect Disord. 2021 Feb 1;280(Pt A):295-304. doi: 10.1016/j.jad.2020.11.030. Epub 2020 Nov 11. PMID 33221715